CLINICAL TRIAL: NCT03712852
Title: Gingival Phenotype Changes After Different Periodontal Plastic Surgical Techniques.
Brief Title: Platelet Rich Fibrin vs Sub Epithelial Connective Tissue and Coronally Advanced Flap Alone in Gingival Recession
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: G. d'Annunzio University (Other)
Responsible Party: Principal Investigator, Michele Paolantonio, professor and chairman, G. d'Annunzio University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 16102018
Record Dates: First submitted 2018-10-16; First posted 2018-10-19 (Actual); Results first posted 2021-02-10 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Gingival Recession
Keywords: Platelet-Rich fibrin; Plastic surgery; Phenotype
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Intervention Model Description: parallel assignment
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PRF+CAF treated patients (Active Comparator): The clot collected from the blood samples is pressed through a calibrated compression system into the PRF box the folded membrane is measured and adjusted to 1,5 mm, then transferred on a sterile gauze. A modified coronally advanced flap technique (MCAF) is used to treat the recession defect, the PRFs are placed over the exposed root surface, ﬂap is coronally positioned and sutures over the enamel in a tension-free position.
  Interventions: Procedure: PRF+CAF treated patients
- SCTG+ CAF treated patients (Active Comparator): SCTG is taken from the opposite palate area of gingival defect. The graft is collected with a single incision technique and it is measured and adjusted to 1,5 mm by measuring with a standard caliper.A modified coronally advanced flap technique (MCAF) is used to treat the recession defect, the SCTGs are placed over the exposed root surface, ﬂap is coronally positioned and sutures over the enamel in a tension-free position.
  Interventions: Procedure: SCTG+ CAF treated patients
- CAF treated patients (Active Comparator): A modified coronally advanced flap technique (MCAF) is used to treat the recession defect, the flap is sutured over the enamel in a tension free position.
  Interventions: Procedure: CAF treated patients

INTERVENTIONS:
Procedure: PRF+CAF treated patients — Patients will be treated by coronally advanced flap with addition of PRF membrane
  Arms: PRF+CAF treated patients
Procedure: SCTG+ CAF treated patients — Patients will be treated by coronally advanced flap with addition of SCTG graft
  Arms: SCTG+ CAF treated patients
Procedure: CAF treated patients — Patients will be treated by coronally advanced flap
  Arms: CAF treated patients

SUMMARY:
Gingival thickness plays a key role not only in the etiology but also in the treatment of gingival recessions. a thin marginal tissue lining the hard periodontal tissues seems to be one of the main risk factor for the onset of gingival recession ; more recently, authors reported that as the gingival thickness decreases, the gingival recession severity increases . When gingival inflammation occurs, if the tissue is thin the consequent destruction can quickly produce a gingival recession (GR) .

When treating a gingival recession, the clinician should aim not only to completely cover the exposed root surface but also to prevent a future recession recurrence Currently, CAF associated with graft is considered as the gold standard for exposed root coverage; this technique has demonstrated high rates in gingival recession reduction and positive predictability in obtaining complete root coverage . However, some disadvantages about this surgical approach can be easily highlighted: patients experience more discomfort, longer chair-time it's necessary and a second wound area is created . On the other hand, CAF procedure alone does not require a second surgical site, with better post-operative course, also reducing the surgical time. However, long term-studies report lower probability of complete root coverage when using the CAF technique without a simultaneous increase of the gingival thickness as compared to CAF+graft treatment.

In this scenario, The Platelet rich fibrin (PRF) could be a valuable alternative treatment of gingival defects. It's a platelet concentrate, obtained by a fast and simple procedure that does not require anticoagulant and bovine thrombin . It can also be categorized as a live tissue thanks to platelets, leukocytes, growth factors and stem cells trapped in a polymerized fibrin mesh. PRF is used in various fields of regenerative medicine; It promotes stabilization and revascularization of the flaps, contributes to soft tissue wound healing and reduces post-operative discomfort.

The purpose of this clinical study will be to determine if the combination of platelet rich fibrine membrane with a modified coronally advanced flap (MCAF) improved the gingival biotype compared to CAF + graft or CAF alone.

DETAILED DESCRIPTION:
This prospective, randomized and controlled clinical trial will compare three modalities of treatment of Miller's class I-II recession: CAF with PRF versus CAF with Sub-epithelial tissue graft (SCTG) versus CAF. From each patient a single recession on a single tooth located in the upper arches will be selected. Clinical parameters will be evaluated at base-line and after 6 months.

The protocol is approved by the "G. D'Annunzio" University Ethical Committee. This study is in accordance with the Declaration of Helsinki of 1975. Patients will be recruited from the Unit of Periodontology, Department of Medical, Oral and Biotechnological Sciences, "G. D'Annunzio" University of Chieti-Pescara, Italy. All the volunteer candidates will sign a written informed consent.

The trial director will be responsible for randomly assigning patients to treatment after enrollment and will not involve with the clinical interventions or the study measurements. A computer-generated table will be used to make the random assignment, known only to the trial director. An opaque envelope will conceal group allocation and will be opened just before the intervention surgery. Matching between group and treatment will be performed by a figure extraneous to the experimentation, responsible even for keeping and breaking the blinding, and known only to him.

Patients and examiners will be masked to group membership; clinical examiners will be blinded to each other. The study analyst will be also blind to group membership. The analyst will receive the data by groups labeled as A and B. The blind will not be broken until after study completion.

At baseline and 6 months after surgery, the following clinical measurements will be recorded on the mid-buccal point of exposed root surface: Gingival thickness (GT) will be determined using a stent at a mid-buccal location about 1 mm apical to the pocket depth (PD) level with a #15 endodontic reamer with a silicon disk stop. The soft tissue will be gently pierced at a 90° angle, until hard tissue will be felt. Once the silicon disk will be in contact with the soft tissue surface, it will be fixed by a drop of cyanoacrylate adhesive. After the careful removal of the reamer, the distance between the reamer tip and the stop will be measured with a calliper accurate to the nearest 0.1 mm. The other measurements will be taken with a periodontal probe and will be recorded to the nearest millimetre as follows: Gingival recession (GR) will be measured as the distance from the cement-enamel junction (CEJ) to the mid-buccal point of the gingival margin. PD and Clinical attachment level (CAL) will be measured as the distance between the bottom of the pocket and the gingival margin and CEJ, respectively. Keratinized tissue (KT) will be recorded from the mid-buccal point of the gingival margin to the mucogingival junction.

Patient morbidity will be evaluated with a visual analogue scale (VAS). Root coverage esthetic score (RES) (Cairo et al., 2009) will be used for assessing aesthetic outcomes of root coverage procedures.

All clinical parameters will be measured by the same investigator. To avoid a calibration probing bias, 60 recession defects will be measured twice within 72 hours. When 90% of the measurements of Gingival thickness will be within 0.3 mm and within 0.5 mm for measurements of GR , calibration will be successfully accepted.

30 ml of blood samples will be collected in 10-ml tubes without anticoagulant and promptly centrifuged at 3,000 revolutions per minute for 10 minutes. The acellular plasma formed in the upper layer will be washed out. The clot, positioned in the middle of the vial, will be cut off from the lower red corpuscles part. Each PRF clot will be folded onto itself in order to double the thickness, and two membranes placed one over the other (quadruple L-PRF layer) represented the L-PRF graft.

The connective tissue graft will be harvested from the palatal area on the opposite side of the gingival defect according to Zucchelli et al12. Briefly, two horizontal and two vertical incisions will delimitate the donor area. The graft will be separated from the underlying tissues by the scalpel's blade oriented parallel to the palatal surface to obtain an about 2 mm thick graft. Then, the graft will be de-epithelialized by a 15c blade and the fatty tissue will be eliminated until obtaining a graft with a thickness of about 1,5 mm. measured by a standard caliper.

Exposed and intrasulcular root surface will be accurately scaled using curettes. A modified coronally advanced flap technique (MCAF) will be used to treat the recession defect. The ﬂap will be elevated as follows: an intrasulcular incision will be performed around the selected tooth, the incision moves on contiguous papillae area, avoiding the gingival margin of adjacent teeth. From each side, from coronal to apical, an oblique incision will be carried out. A split-full-split dissection will be undertaken until the CEJ could be passively cover by the flap. Both papillae will be de-epithelialized. The PRFs and the SCTGs will be placed over the exposed root surface of the Test group and Control 1 group respectively. The gingival defect will be fully lined by grafts that mildly cover the neighbouring sub-papillae areas. The grafts will be fixed applying suture to the periosteum below. In each group, ﬂap will be coronally positioned and sutured over the enamel in a tension-free position.

All patients will receive 2 g/day amoxicillin+clavulanic acid for 6 days for post-operative infection prevention; 400 mg of oral ibuprofen, twice daily, will control the pain; 0.12% chlorhexidine rinses, twice daily for 3 weeks, will be prescribe to the patients. Sutures will be removed after 14 days. Only 2-4 weeks after sutures removal, respectively, cautious brushing by a soft toothbrush and interdental brushing will be recommend; meantime, the patients use a 1% chlorhexidine gel twice daily. Weekly supra-gingival professional hygiene and motivational reinforcement will be administer to the patients for 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* a full-mouth plaque score (FMPS)* and a full-mouth bleeding score (FMBS)* lower than 20%, at the time of surgery
* to have at least 20 teeth at leat 1 maxillary tooth exhibiting a single Miller second class of gingival recession .

Exclusion Criteria:

* no systemic diseases;
* no coagulation disorders;
* no medications affecting periodontal status in the previous 6 months;
* no pregnancy or lactation;
* no presence of cervical carious lesions,;
* no periodontal surgery on the experimental sites
* no smoking habits
* no inadequate endodontic treatment at the site of surgery
* no presence of cervical carious lesions

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-10-20 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-07-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- G. d'Annunzio University, Chieti, CH, Italy

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- PRF+CAF Treated Patients: Blood samples are collected in four 10-ml tubes without anticoagulant and promptly centrifuged at 3,000 revolutions per minute for 10 minutes The clot, positioned in the middle of the vial, is cut off from the lower red corpuscles part (Fig). The clot is pressed through a calibrated compression system into the PRF box the folded membrane is transferred on a sterile gauze. A modified coronally advanced flap technique (MCAF) is used to treat the recession defect, the PRFs are placed over the exposed root surface, ﬂap is coronally positioned and sutures over the enamel in a tension-free position.
  PRF+CAF treated patients: Patients will be treated by coronally advanced flap with addition of PRF membrane
- SCTG+ CAF Treated Patients: SCTG is taken from the opposite palate area of gingival defect. The graft is collected with a single incision technique and it is measured and adjusted to 1 mm by measuring with a standard caliper.A modified coronally advanced flap technique (MCAF) is used to treat the recession defect, the SCTGs are placed over the exposed root surface, ﬂap is coronally positioned and sutures over the enamel in a tension-free position.
  SCTG+ CAF treated patients: Patients will be treated by coronally advanced flap with addition of SCTG graft
Period: Overall Study
Arm/Group | PRF+CAF Treated Patients | SCTG+ CAF Treated Patients | CAF Treated Patients
Started | 20 | 20 | 20
Completed | 20 | 20 | 20
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Sixty patients (twenty-seven women), aged 18 to 47 years, (mean 32.4 ± 5.0 years) enroll in this study, after their visit at the Unit of Periodontology of the "G. D'Annunzio" University.
Groups:
- Total: Total of all reporting groups
Arm/Group | PRF+CAF Treated Patients | SCTG+ CAF Treated Patients | CAF Treated Patients | Total
Number analyzed (Participants) | 20 | 20 | 20 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 20 | 60
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.4 (5) | 32.4 (5) | 32.4 (5) | 32.4 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Sex: Female | 9 | 9 | 9 | 27
  Sex: Male | 11 | 11 | 11 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 1 | 5
  Not Hispanic or Latino | 18 | 18 | 19 | 55
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Italy | 20 | 20 | 20 | 60

OUTCOME MEASURES:

1. Primary Outcome: Gingival Thickness
Description: the change from baseline measured as the thickness of keratinized tissue recorded at 1 mm from the gingival margin
Time Frame: baseline and 6 months
Population: Statistical software R 3.5.1 was used to analyze the clinical data. Descriptive statistics of GT was analyzed by non-parametric Cliff's delta tests to asses group dominance and by a Heteroscedastic ANOVA with Games-Howell posthoc tests.
Measure: Mean (Standard Deviation); unit: millimeter
Arm/Group | PRF+CAF Treated Patients | SCTG+ CAF Treated Patients | CAF Treated Patients
Number analyzed (Participants) | 20 | 20 | 20
millimeter | 1.97 (0.55) | 1.95 (0.28) | 1.39 (0.46)
Statistical Analysis 1: Comparison: PRF+CAF Treated Patients vs SCTG+ CAF Treated Patients vs CAF Treated Patients; Test type: Superiority; Mean Difference (Net) = 0.92, 95% CI 2-sided [0.68 to 1.17]; Multiple univariate analyses for each variable were performed. GT was analyzed by non-parametric Cliff's delta tests to assess group dominance and by a Heteroscedastic ANOVA with Games-Howell posthoc tests. A sensitivities analysis with different types of robust analyses (M-estimators and High Breakdown LTS Estimators, both with Huber's, Hampel's and Biweight's loss functions) was conducted to get an effect-size estimate by means of Bootstrap Bias Corrected and accelerated (BCa) 95% Confidence Intervals

2. Secondary Outcome: Gingival Recession
Description: the change from baseline measured as the distance between the cemento enamel junction and the gingival margin
Time Frame: baseline and 6 months
Measure: Mean (Standard Deviation); unit: millimeter
Arm/Group | PRF+CAF Treated Patients | SCTG+ CAF Treated Patients | CAF Treated Patients
Number analyzed (Participants) | 20 | 20 | 20
millimeter | 3.28 (0.59) | 3.70 (0.73) | 3.05 (1.10)
Statistical Analysis 1: Comparison: PRF+CAF Treated Patients vs SCTG+ CAF Treated Patients vs CAF Treated Patients; Test type: Superiority; Median Difference (Final Values) = 3.28, 95% CI 2-sided [3.00 to 3.55]; This outcome was analyzed by posthoc Nemenyi's tests

3. Secondary Outcome: Keratinized Tissue
Description: the change from baseline measured as the distance of the mid-buccal site of the gingival margin to the mucogingival junction
Time Frame: baseline and 6 months
Measure: Mean (Standard Deviation); unit: millimeter
Arm/Group | PRF+CAF Treated Patients | SCTG+ CAF Treated Patients | CAF Treated Patients
Number analyzed (Participants) | 20 | 20 | 20
millimeter | 0.08 (0.25) | 2.00 (0.97) | -0.15 (0.67)
Statistical Analysis 1: Comparison: PRF+CAF Treated Patients vs SCTG+ CAF Treated Patients vs CAF Treated Patients; Test type: Superiority; Mean Difference (Final Values) = 0.08, 95% CI 2-sided [-0.46 to 2.46]; This outcome was analyzed by posthoc Nemenyi's tests

4. Secondary Outcome: Pocket Depth
Description: the change from baseline measured as the distance between the bottom of the pocket and the gingival margin
Time Frame: baseline and 6 months
Measure: Mean (Standard Deviation); unit: millimeter
Arm/Group | PRF+CAF Treated Patients | SCTG+ CAF Treated Patients | CAF Treated Patients
Number analyzed (Participants) | 20 | 20 | 20
millimeter | 0.20 (0.34) | -0.10 (0.64) | 0.45 (0.51)
Statistical Analysis 1: Comparison: PRF+CAF Treated Patients vs SCTG+ CAF Treated Patients vs CAF Treated Patients; Test type: Superiority; Mean Difference (Final Values) = 0.20, 95% CI 2-sided [-0.40 to 0.69]; This outcome was analyzed by posthoc Nemenyi's tests

5. Secondary Outcome: Clinical Attachment Level
Description: the change from baseline measured as the distance between the bottom of the pocket and the CEJ
Time Frame: baseline and 6 months
Measure: Mean (Standard Deviation); unit: millimeter
Arm/Group | PRF+CAF Treated Patients | SCTG+ CAF Treated Patients | CAF Treated Patients
Number analyzed (Participants) | 20 | 20 | 20
millimeter | 3.38 (0.89) | 3.60 (0.60) | 3.40 (0.89)
Statistical Analysis 1: Comparison: PRF+CAF Treated Patients vs SCTG+ CAF Treated Patients vs CAF Treated Patients; Test type: Superiority; Mean Difference (Final Values) = 3.38, 95% CI 2-sided [2.96 to 3.81]; CAL was analyzed with both Nemenyi's tests and a Moderated Regression (Treatment by Baseline values)

6. Secondary Outcome: Patient Reported Outcomes (PROMs)
Description: A visual analogical scale (VAS) will be used to assess the patient morbidity after treatment. The scale has 10 numerical values, from 1(better outcome) to 10 (worse outcome).
Time Frame: 2 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | PRF+CAF Treated Patients | SCTG+ CAF Treated Patients | CAF Treated Patients
Number analyzed (Participants) | 20 | 20 | 20
score on a scale | 3.37 (0.326) | 3.58 (0.322) | 4.73 (0.343)

7. Secondary Outcome: Aesthetic
Description: Aesthetic outcome will be recorded using the root coverage esthetic score (RES) introduced by Cairo et al. in 2009. This score assess five domains: level of the gingival margin, marginal tissue contour, soft tissue texture, mucogingival junction alignment, and gingival color. Zero, 3, or 6 points will be used for the evaluation of the position of the gingival margin, whereas a score of 0 or 1 point will be used for each of the other variables.The value assigned for root coverage will be 60% of the total score, whereas 40% will be assigned to the other four variables. 3 points will be given for partial root coverage, and 6 points will be given for complete root coverage; 0 points will be assigned when the final position of the gingival margin is equal or apical to the previous recession. One point will be assigned for each of the other four variables. Thus, 10 points will be a perfect score. 0-10 higher score indicates better outcome.
Time Frame: 6 months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | PRF+CAF Treated Patients | SCTG+ CAF Treated Patients | CAF Treated Patients
Number analyzed (Participants) | 20 | 20 | 20
units on a scale | 2.56 (0.222) | 2.50 (0.230) | 2.74 (0.240)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | PRF+CAF Treated Patients | SCTG+ CAF Treated Patients | CAF Treated Patients
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-08): https://cdn.clinicaltrials.gov/large-docs/52/NCT03712852/Prot_SAP_000.pdf